CLINICAL TRIAL: NCT01141114
Title: Randomized Controlled Trial of Patient Navigation to Increase Colorectal Cancer Screening Rates Among Community Health Center Patients
Brief Title: Study of Patient Navigation to Promote Colon Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: American Cancer Society, Inc. (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MRSGT-05-007-01-CPPB
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer Screening
Keywords: community health centers; colorectal cancer screening; urban health
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of a Patient Navigator (Experimental)
  Interventions: Other: Patient navigation
- Usual Care (Other): No Intervention - usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Patient navigation — Letter and Colorectal Cancer Screening Brochure mailed to patients. Telephone outreach by Patient Navigators.
  Arms: Use of a Patient Navigator
Other: Usual care — Usual care
  Arms: Usual Care

SUMMARY:
This study will investigate whether patient navigation can increase rates of colorectal cancer screening among linguistically and culturally diverse disadvantaged patients served by urban community health centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 52-75 who had one visit to a primary care physician in a community health center in each of the 2 previous years and who have not received colorectal cancer screening based on HEDIS criteria.

Exclusion Criteria:

* Current cancer diagnosis, undergoing treatment (or treatment completed within the past year)
* Severe cardiac disease (high-risk CAD,9 valvular disease, NYHA Class III or IV CHF, EF < 35%)
* Severe COPD (FEV1< 1liter or on home oxygen)
* CVA with severe functional impairment (aphasia or hemiparesis)
* MS with severe functional impairment
* Renal failure with CrCl< 30 or on dialysis
* Gastrointestinal symptoms (pain, bleeding, etc) within the past 6 months
* Chronic active liver disease or cirrhosis, with albumin < 3 or elevated INR
* Advanced HIV disease (CD4 count <200)
* Severe lupus (with cerebritis or renal failure as defined above)
* Severe complications of diabetes (blindness, amputations other than toes)
* Advanced Dementia
* Psychosis
* Paranoia
* Active substance abuse
* Schizophrenia
* Psychiatric hospitalization within the past year

Ages: 52 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
completion of colorectal cancer screening | 1 year

SECONDARY OUTCOMES:
Comparison of detection of polyps and cancers in intervention vs. control groups | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Lasser, MD, MPH, Principal Investigator — Cambridge Health Alliance/Harvard Medical School
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Lasser KE, Ayanian JZ, Fletcher RH, Good MJ. Barriers to colorectal cancer screening in community health centers: a qualitative study. BMC Fam Pract. 2008 Feb 27;9:15. doi: 10.1186/1471-2296-9-15. PMID 18304342
- [Derived] Lasser KE, Murillo J, Lisboa S, Casimir AN, Valley-Shah L, Emmons KM, Fletcher RH, Ayanian JZ. Colorectal cancer screening among ethnically diverse, low-income patients: a randomized controlled trial. Arch Intern Med. 2011 May 23;171(10):906-12. doi: 10.1001/archinternmed.2011.201. PMID 21606094